CLINICAL TRIAL: NCT05692557
Title: Role of Virtual Reality Distraction Technique to Improve Chest Burns With Acute Respiratory Distress Syndrome (ARDS) Following Smoke Inhalation in Community-dwelling Middle-aged Adults - A Randomized Controlled Study.
Brief Title: Virtual Reality Distraction Technique to Improve Chest Burns With Acute Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Associate Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHPT/020/087
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Burns Chest Left Lateral; Burns Chest Right Lateral; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: This trial was a randomized, parallel-group, clinical controlled trial conducted at the department of health and rehabilitation sciences, college of applied medical sciences, Prince Sattam bin Abdulaziz University, Al Kharj, Saudi Arabia.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants were not aware of which treatment they were receiving (blind participants); however, they were informed that they would receive one of the two interventions. Due to the nature of the interventions, it was not possible to blind the therapist who treated the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality distraction and chest physiotherapy (Experimental): Virtual reality distraction: The Oculus Rift's "Fujii - Mystical Journey" was a game played by the Virtual reality distraction group on a tablet. The game is a peaceful, ethereal voyage that passes through several surreal, natural locations. The game combines elements of adventure, agriculture and revitalizing music. It alternates between outdoor exploration and inventive gardening. Players explore three different magical biomes. The life force in each biome is restored by interacting with the plants and animals there. Before beginning the chest physical therapy, the patients had 15 minutes to play this computer game
  Interventions: Device: Virtual reality
- Progressive relaxation exercise and chest physiotherapy (Active Comparator): Progressive muscle relaxation: The patients of the control group performed the Progressive muscle relaxation technique, a relaxation technique used to control pain. It is believed that anxiety-inducing thoughts result in muscle tension and hence muscle relaxation can reduce anxiety. The relaxation technique consisted of tensing and relaxing different muscles, starting from the toes and finally involving muscles of the head and neck. It was recommended that this be done in a peaceful, distraction-free environment. The muscle groups were tensed for a period of 5 seconds and then relaxed for 30 seconds, the process was repeated for a period of 15 minutes
  Interventions: Procedure: Progressive muscle relaxation

INTERVENTIONS:
Device: Virtual reality — The Oculus Rift's (Lenovo, Beijing, China) "Fujii - Mystical Journey" was the game played by the VRD group on a tablet. The game is a peaceful, ethereal voyage that passes through several surreal, natural locations.
  The game combines elements of adventure, agriculture and revitalizing music. It alternates between outdoor exploration and inventive gardening. Players explore three different magical biomes. The life force in each biome is restored by interacting with the plants and animals there.
  Arms: Virtual reality distraction and chest physiotherapy
Procedure: Progressive muscle relaxation — The patients of the control group performed Progressive muscle relaxation technique, a relaxation technique used to control pain. It is believed that anxiety-inducing thoughts result in muscle tension and hence muscle relaxation can reduce anxiety. The relaxation technique consisted of tensing and relaxing different muscles, starting from the toes and finally involving muscles of the head and neck. It was recommended that this be done in a peaceful, distraction-free environment. The muscle groups were tensed for a period of 5 seconds and then relaxed for 30 seconds.
  Arms: Progressive relaxation exercise and chest physiotherapy

SUMMARY:
Inhalation of toxic gases and chemical irritants during the fire leads to damage to the respiratory tract or the alveolar tissue, which is known as smoke inhalation injury. Acute Respiratory Distress Syndrome (ARDS) is associated with smoke inhalation injury. These patients usually need physiotherapy in the form of chest mobilization and breathing exercises for up to 4 to 6 weeks after discharge from the burns care centre. The patients during this phase are usually in pain and extremely anxious about these exercises. Virtual reality distraction (VRD) is one such technique that is gaining immense popularity recently, it has more immersive distraction when compared to traditional distraction techniques. This study aims to investigate the effect of a virtual reality distraction (VRD) technique as a pain alleviation tool for reducing pain during physiotherapy in burns patients with acute respiratory distress syndrome (ARDS) in a hospital setting.

DETAILED DESCRIPTION:
Burns of the chest region (Chest burns - CB) constitute a common burn (29%) among other types of burn, in which second and third-degree burns are the most common type of injuries noted. Additionally, inhalation of toxic gases and chemical irritants during the fire leads to damage to the respiratory tract or the alveolar tissue, which is known as smoke inhalation injury. Acute Respiratory Distress Syndrome (ARDS) is associated with smoke inhalation injury, which is one of the infectious complications after a burn injury. According to the present data, the incidence of ARDS in burn patients is about 20 - 56% and is one of the main causes of death among burn patients. Management of ARDS generally includes mechanical ventilation, prophylaxis treatment, proper diet and physiotherapy treatment. These patients usually need physiotherapy in the form of chest mobilization and breathing exercises for up to 4 to 6 weeks after discharge from the burns care centre. The patients during this phase are usually in pain and extremely anxious about these exercises, hence pain and anti-anxiety drugs may be prescribed. Virtual reality distraction (VRD) is one such technique that is gaining immense popularity recently, it has more immersive distraction when compared to traditional distraction techniques like inhibition exercises, meditation or progressive muscle relaxation exercises. This study aims to investigate the effect of a virtual reality distraction (VRD) technique as a pain alleviation tool for reducing pain during physiotherapy in burns patients with acute respiratory distress syndrome (ARDS) in a hospital setting.

ELIGIBILITY:
Inclusion Criteria:

Community-dwelling middle-aged adult patients (aged between 35 - 55 years) with chest burn injury and moderate ARDS who were to receive physiotherapy at home for at least 1 month were invited to participate. The clinical diagnosis of ARDS (International Classiﬁcation of Diseases 10th revision [ICD-10] group J80) was diagnosed according to Berlin diagnostic criteria by a general physician. The baseline pain intensities 3 to 8 on the visual analogue scale (VAS) were included.

Exclusion Criteria:

Any injury that would hinder the outcome of the study procedures, patients who had difficulty in communication due to impaired hearing, visual or motor development, who had a history of epilepsy, migraine or motion sickness, and participants who were suspected victims of abuse.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity - Visual analog scale (VAS) | Baseline
  The participants were asked to mark their level of pain intensity between 0 and 10, in which '0' denotes "no pain at all" and '10' denotes "the worst pain ever possible". It is a reliable and valid tool to assess pain intensity as proven by studies and a 2-point change or response in the NPRS is considered a clinically meaningful change that exceeds measurement error.
Pain intensity - Visual analog scale (VAS) | 4 weeks
  The participants were asked to mark their level of pain intensity between 0 and 10, in which '0' denotes "no pain at all" and '10' denotes "the worst pain ever possible". It is a reliable and valid tool to assess pain intensity as proven by studies and a 2-point change or response in the NPRS is considered a clinically meaningful change that exceeds measurement error.
Pain intensity - Visual analog scale (VAS) | 8 weeks
  The participants were asked to mark their level of pain intensity between 0 and 10, in which '0' denotes "no pain at all" and '10' denotes "the worst pain ever possible". It is a reliable and valid tool to assess pain intensity as proven by studies and a 2-point change or response in the NPRS is considered a clinically meaningful change that exceeds measurement error.
Pain intensity - Visual analog scale (VAS) | 6 months
  The participants were asked to mark their level of pain intensity between 0 and 10, in which '0' denotes "no pain at all" and '10' denotes "the worst pain ever possible". It is a reliable and valid tool to assess pain intensity as proven by studies and a 2-point change or response in the NPRS is considered a clinically meaningful change that exceeds measurement error.

SECONDARY OUTCOMES:
Pulmonary function test - forced vital capacity (FVC) | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - forced vital capacity (FVC) | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - forced vital capacity (FVC) | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - forced vital capacity (FVC) | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - forced expiratory volume in 1 second (FEV1) | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - forced expiratory volume in 1 second (FEV1) | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - forced expiratory volume in 1 second (FEV1) | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - forced expiratory volume in 1 second (FEV1) | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - FEV1/FVC | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - FEV1/FVC | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - FEV1/FVC | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - FEV1/FVC | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - peak expiratory flow (PEF) | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - peak expiratory flow (PEF) | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - peak expiratory flow (PEF) | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - peak expiratory flow (PEF) | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - residual volume (RV) | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - residual volume (RV) | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - residual volume (RV) | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - residual volume (RV) | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - functional residual capacity (FRC) | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - functional residual capacity (FRC) | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - functional residual capacity (FRC) | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - functional residual capacity (FRC) | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - total lung capacity (TLC) | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - total lung capacity (TLC) | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - total lung capacity (TLC) | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - total lung capacity (TLC) | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - RV/TLC | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - RV/TLC | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - RV/TLC | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - RV/TLC | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - diffusing capacity for carbon monoxide of the lungs (DLCO) | Baseline
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - diffusing capacity for carbon monoxide of the lungs (DLCO) | 4 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - diffusing capacity for carbon monoxide of the lungs (DLCO) | 8 weeks
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.
Pulmonary function test - diffusing capacity for carbon monoxide of the lungs (DLCO) | 6 months
  Pulmonary function test (PFT) was undertaken to determine the degree of functional impairment and was performed with spirometer (MasterScreen Body; Jaeger, Wurzburg, Germany). The lung functions were determined by blowing through the mouth piece in the spirometer. The test was repeated three times or more and average score was considered, and all values were expressed as a percentage of the predicted values.

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Nambi, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Dr. Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The study will be published in the impacted journal.